CLINICAL TRIAL: NCT05995496
Title: Dynamic Neural Computations Underlying Cognitive Control in Bulimia Nervosa
Brief Title: Changes in Inhibition and Valuation After Eating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laura Berner, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY-22-01587; 1R01MH132786 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Bulimia Nervosa
MeSH Terms: conditions — Bulimia Nervosa | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Two participant groups (one with and one without bulimia nervosa) will be scanned using MRI after they have fasted and after they have consumed a standardized meal. The order of these two scans will be counterbalanced across groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with Bulimia Nervosa (Experimental): Participants are randomly assigned (in even numbers across the two groups) to scan order:
  A. These participants are first scanned after 16 hours of fasting on one day, and are next scanned after a standardized meal on a second day.
  B. These participants are first scanned after a standardized meal on one day, and are next scanned after 16 hours of fasting on a second day.
  Interventions: Other: Fasting state; Other: Fed state; Other: Magnetic Resonance Imaging
- Participants without Bulimia Nervosa (Active Comparator): Participants are randomly assigned (in even numbers across the two groups) to scan order:
  A. These participants are first scanned after 16 hours of fasting on one day, and are next scanned after a standardized meal on a second day.
  B. These participants are first scanned after a standardized meal on one day, and are next scanned after 16 hours of fasting on a second day.
  Interventions: Other: Fasting state; Other: Fed state; Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Fasting state — 16 hours of fasting
Other: Fed state — Fed a standardized meal
Other: Magnetic Resonance Imaging — Neuroimaging with computational modeling
  Other Names: MRI

SUMMARY:
An impaired ability to exert control has been implicated in bulimia nervosa (BN), but this impairment may not represent a stable trait or be the most effective focus for treatment. This project aims to understand how predictions and value-based decisions about control may be abnormally influenced by eating in individuals with BN, thereby maintaining cycles of binge eating, purging, and restriction.

DETAILED DESCRIPTION:
The overarching goal of this project is to test a neurocomputational model of BN that incorporates learning and decision-making components of control. The study combines functional magnetic resonance imaging (fMRI), computational modeling, and real-time mobile assessments to examine the influences of acute fasting and eating on brain function and associated control-related updating and effort-valuation processes in BN. More specifically, the study has the following main objectives: 1) To determine the influence of eating on control-related prediction updating in BN.; 2) To determine the influence of eating on control-related cognitive effort valuation in BN; 3) To use state-specific neural activation to predict BN symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 to 45 years
* Current BMI greater than or equal to 18.5kg/m2 but under 30kg/m2
* Right-handed
* English-speaking

Additional Inclusion Criteria for Women with Bulimia Nervosa:

* Meet DSM-5 criteria for bulimia nervosa

Exclusion Criteria:

* Medical instability
* Ongoing medical treatment, medical condition, or psychiatric disorder that may interfere with study variables or participation
* Shift work
* Pregnancy, planned pregnancy, or lactation during the study period
* Allergy to any of the ingredients in or unwillingness to consume the standardized meal or unwillingness to drink water during the fasting period
* Any contraindication for fMRI

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The prevalence of bulimia nervosa is substantially greater in women than in men. Moreover, prior research suggest that men and women show different neural response patterns during the engagement of inhibitory control, and that satiety differentially impacts the neural function of men and women.
Enrollment: 150 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Frontostriatal Activation Associated with Prediction Errors on the Stop Signal Task | 1-2.5 hours after a 16-hour fast (fasted state)
  Blood oxygen level dependent (BOLD) signal in frontostriatal brain circuitry associated with inhibitory control prediction errors
Frontostriatal Activation Associated with Prediction Errors on the Stop Signal Task | 1-2.5 hours after a standardized meal (fed state)
  Blood oxygen level dependent (BOLD) signal in frontostriatal brain circuitry associated with inhibitory control prediction errors
Frontostriatal Activation Encoding the Subjective Value of Cognitive Effort on the Cognitive-Effort Discounting Task | 1-2.5 hours after a 16-hour fast (fasted state)
  Blood oxygen level dependent (BOLD) signal in frontostriatal brain circuitry associated with the subjective value of expending cognitive effort on control
Frontostriatal Activation Encoding the Subjective Value of Cognitive Effort on the Cognitive-Effort Discounting Task | 1-2.5 hours after a standardized meal (fed state)
  Blood oxygen level dependent (BOLD) signal in frontostriatal brain circuitry associated with the subjective value of expending cognitive effort on control

SECONDARY OUTCOMES:
Percent correct responses to stop trials and the trial-by-trial association | 1-2.5 hours after a 16-hour fast (fasted state)
  Behavioral performance on the stop signal task, as measured by percent correct responses to stop trials and the trial-by-trial association between the predicted likelihood that upcoming inhibition is needed (P(stop)) from a Bayesian ideal observer model and accuracy
Percent correct responses to stop trials and the trial-by-trial association | 1-2.5 hours after a standardized meal (fed state)
  Behavioral performance on the stop signal task, as measured by percent correct responses to stop trials and the trial-by-trial association between the predicted likelihood that upcoming inhibition is needed (P(stop)) from a Bayesian ideal observer model and accuracy
Cognitive Effort Discounting Task Behavioral Performance | 1-2.5 hours after a 16-hour fast (fasted state)
  The subjective value of cognitive effort estimated for each N-back load level and cost- and benefit-modulated drift rate parameters from a drift- diffusion model applied to behavioral performance data
Cognitive Effort Discounting Task Behavioral Performance | 1-2.5 hours after a standardized meal (fed state)
  The subjective value of cognitive effort estimated for each N-back load level and cost- and benefit-modulated drift rate parameters from a drift- diffusion model applied to behavioral performance data
Binge-eating Severity | Baseline and 6-month follow-up
  The frequency of binge-eating episodes as assessed by the Eating Disorder Examination (EDE) and Ecological Momentary Assessment (EMA). Binge-eating frequency has a minimum limit of 0 and no maximum limit. A higher score indicates a greater severity.
Compensatory Behavior Severity | Baseline and 6-month follow-up
  The frequency of compensatory behaviors as assessed by the EDE and EMA. This frequency has a minimum limit of 0 and no maximum limit. A higher score indicates a greater severity.
Dietary Restriction Severity | Baseline and 6-month follow-up
  The frequency of fasting episodes as assessed by the EDE avoidance of eating item (minimum limit = 0, maximum limit = 6); the severity of dietary restriction as assessed by the Eating Pathology Symptoms Inventory (EPSI) - restricting subscale (minimum limit=0; maximum limit=24), and the frequency of restrictive eating behaviors as assessed by EMA (minimum limit=0; no maximum limit). On all measures, a higher score indicates a greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Berner, Ph.D., Principal Investigator — Mount Sinai Icahn School of Medicine
Locations (1):
- Center of Excellence in Eating and Weight Disorders at the Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Specify Other Time FrameWithin one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Specify Other Mechanism All data will be deposited to the National Data Archive (NDA) starting 12 months after the award begins and will be deposited every 6 months thereafter following the usual NDA data submission dates. The research community will be able to find the data through this study's NDA Collection C4723. The research community will have access to the data within one year of the completion of the funded project period or upon acceptance of the data for publication, whichever is earlier. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
URL: https://nda.nih.gov/edit_collection.html?id=4723